CLINICAL TRIAL: NCT04909593
Title: Study to Evaluate Automated Intensity Management in Patients Undergoing a BSC SCS Temporary Trial: The AIM Study
Brief Title: Study to Evaluate Automated Intensity Management in Patients Undergoing a BSC SCS Temporary Trial
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4091
Record Dates: First submitted 2021-05-21; First posted 2021-06-02 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain; Intractable Pain; Low Back Pain; Pain, Neuropathic; Pain, Back
MeSH Terms: conditions — Chronic Pain; Pain, Intractable; Low Back Pain; Neuralgia; Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Spinal Cord Stimulation (Experimental): SCS trial systems including external trial stimulators, lead(s)/extensions(s), and operating room (OR) cable(s)/extender(s) and optional sensor.
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Spinal cord stimulation at varied electrode, pulse width, frequency and amplitude parameters
  Other Names: neurostimulation

SUMMARY:
The purpose of the study is to assess the feasibility of using information extracted from physiologic signals to automatically adjust stimulation in patients undergoing Spinal Cord Stimulation (SCS).

ELIGIBILITY:
Key Inclusion Criteria:

* Study candidate is undergoing a temporary SCS trial of commercially approved BSC neurostimulator system, per local directions for use (DFU).
* Subject signed a valid, EC/IRB-approved informed consent form.
* Age 18 or above, or above legal age and willing and capable of giving informed consent specific to national law when written informed consent is obtained.
* In the clinician best judgment, subject is able to distinguishably describe quality and location of sensation and pain.

Key Exclusion Criteria:

* Subject meets any contraindication in BSC neurostimulation system local DFU.
* Investigator-suspected gross lead migration during the SCS trial period which may preclude the study candidate from receiving adequate SCS therapy.
* Subject is currently diagnosed with cognitive impairment, or exhibits any characteristic, that in the clinician's best judgement would limit study candidate's ability to assess and report sensation information.
* Subject is currently diagnosed with a physical impairment, or exhibits a condition that would limit study candidate's ability to complete study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (1):
- PCPMG Clinical Research Unit, LLC, Greenville, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spinal Cord Stimulation
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All consented subjects
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17
  Native American | 1
  Black, of African Heritage | 2
  American Indian or Alaska Native | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Perception Threshold
Description: Percent change in patient's perceiving spinal cord stimulation (i.e. Perception Threshold) when going from a reclining to sitting position in a reclining chair
Time Frame: Programming Visit (up to 15 days post-screening)
Population: Subjects who received programming with SCS trial neurostimulator system.
Measure: Mean (Standard Deviation); unit: percent change in perception threshold
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 20
percent change in perception threshold | 157 (52)

ADVERSE EVENTS:
Time Frame: From Informed consent through End of Study Visit (approximately 15 days).
Description: Other (Not including Serious) Adverse Events reported include device hardware and/or procedure related adverse events which were monitored/assessed.
  All Serious Adverse Events and All-Cause Mortality were monitored/assessed.
Arm/Group | Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04909593/Prot_002.pdf